CLINICAL TRIAL: NCT03493061
Title: Systemic Chemotherapy With Irinotecan Plus Hepatic Arterial Infusion With Floxuridine and Oxaliplatin in Patients With Initially Unresectable Colorectal Liver Metastasis: A Prospective Study
Brief Title: A Study of Systemic Chemotherapy With CPT-11 Plus HAI (FUDR+L-OHP) in Patients With Initially Unresectable CRCLM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Yuhong Li, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAI-CRCLM
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Colo-rectal Cancer; Liver Metastases
MeSH Terms: conditions — Colonic Neoplasms | interventions — Irinotecan; Oxaliplatin; Floxuridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic CPT-11 + HAI (FUDR+L-OHP) (Experimental): Patients will receive Systemic CPT-11 + HAI (FUDR+L-OHP) every 28 days:
  Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; followed by Oxaliplatin 85 mg/m2 over 3 hours through the HAI pump on Day 1 and 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.
  then Irinotecan 150 mg/m2 IV over 90 minutes on Day 15, followed by Oxaliplatin 85 mg/m2 IV over 3 hours on Day 15.
  This will be repeated on Day 1 of each 28-day cycle. FUDR will be administered through a 14-day continuous infusion with the HAI pump.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Floxuridine

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 150 mg/m2 IV over 90 minutes on Day 1, 15
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 over 3 hours will be administered through the HAI pump on day 1. Oxaliplatin 85 mg/m2 IV over 3 hours on day 15.
Drug: Floxuridine — 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.

SUMMARY:
The aim of the trial is to optimize response rates and rates of secondary resections of metastases in patients with initially non-resectable metastatic colorectal cancer Liver Metastasis. The patients will be treated with systemic chemotherapy With irinotecan plus hepatic arterial infusion With floxuridine and oxaliplatin

DETAILED DESCRIPTION:
Recent studies and our experience have proved the efficacy and safety of systemic chemotherapy combined with hepatic arterial infusion (HAI) with floxuridine and dexamethasone in patients with initially unresectable colorectal liver metastasis. Hepatic arterial infusion oxaliplatin trials have been done with oxaliplatin alone and in combination with irinotecan, 5-FU/LV, and mitomycin-C and have showed that Hepatic arterial infusion oxaliplatin could increase response rate and resection rate for colorectal liver metastasis. Therefore, we designed this study to determine whether systemic chemotherapy With irinotecan plus hepatic arterial infusion With floxuridine and oxaliplatin can increase the complete resection rate (R0) and improve the overall survival in patients with initially unresectable colorectal liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old
* Histologically confirmed colorectal adenocarcinoma
* Radiologically or pathologically confirmed diagnosis of colorectal liver metastasis
* Initially unresectable colorectal liver metastasis confirmed by the multidisciplinary team (MDT)
* With no prior treatment for liver metastasis, including chemotherapy, operation, radiotherapy, transcatheter hepatic arterial chemoembolization (TACE) and targeted therapy
* Without extra-hepatic metastasis confirmed by CT, MRI or PET/CT (if necessary) scanning
* With adequate bone marrow function: platelets ≥ 90 x 109/L; white blood cells ≥ 3×109/L; absolute neutrophil count (ANC) ≥ 1.5 x 109/L Serum bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 5 x ULN
* Patient has no ascites and with adequate blood coagulation function, albumin ≥ 35 g/L
* Grade A level of Child-Push Liver Function
* Creatinine ≤ 1× ULN, or Calculated Creatinine Clearance >50ml/min （Cockcroft-Gault Equation）
* ECOG performance status of 0-2
* Life expectancy ≥ 3 months
* Not appropriate for anti-EGFR or any other targeted therapy (with KRAS mutation or could not afford it)
* Patients have provided a signed Informed Consent Form
* With good compliance

Exclusion Criteria:

* With any extra-hepatic metastasis and/or primary tumor recurrence
* Severe arterial embolism or ascites
* With hemorrhagic tendency or coagulation disorders
* Hypertensive crisis or hypertensive encephalopathy
* Severe and uncontrolled systemic complications such as infections or diabetes.
* Serious cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), uncontrolled hypertension even with appropriate drug intervention, unstable angina pectoris, congestive heart failure (NYHA 2-4 degree), arrhythmia that needs medication intervention
* Patient who has suffered from central nervous system diseases such as primary brain tumor, uncontrolled epilepsy even with standard treatment, any brain metastasis or stroke
* Patient who has a concurrent malignancy or has a malignancy within 5 years before study enrollment, (with the exception of radically resected skin basal cell carcinoma or cervical carcinoma in situ)
* Patient who has received any investigational antineoplastic agent within 28 days before the enrollment
* Any residual toxicity from prior chemotherapy (with the exception of alopecia), such as grade 2 or more sensory peripheral neuropathy (NCI CTC v3.0), oxaliplatin-based regimen will not be considered
* Patient who is allergic to oxaliplatin, leucovorin, 5-Fluorouracil, floxuridine or dexamethasone
* Pregnant or lactating women
* Patient who does not use or refuses to take any appropriate contraceptive measures (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or sterilization operation), including women of childbearing age (within 2 years after the last menstrual period) and men who are with possible fertility
* Unable or unwilling to comply with the research plan
* The existence of any other disease, dysfunction caused by metastatic lesions, or suspicious disease found on the regular examination, which indicating contraindications to the use of study drugs or may bring high risks of treatment related complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Complete resection rates (R0 resection rates) | Up to 2-4 months
  defined as no macroscopic or microscopic residual tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol